CLINICAL TRIAL: NCT00305084
Title: A Phase IB Study of NGR-hTNF in Combination With Doxorubicin in Patients Affected by Advanced or Metastatic Solid Tumors
Brief Title: Study of NGR-hTNF in Combination With Doxorubicin in Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AGC Biologics S.p.A. (Industry)
Responsible Party: Molmed, Molmed
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NGR003; EUDRACT Number: 2005-004846-15
Record Dates: First submitted 2006-03-15; First posted 2006-03-21 (Estimated); Results first posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-09

CONDITIONS: Cancer
Keywords: NGR-hTNF; doxorubicin; solid tumors
MeSH Terms: conditions — Neoplasms | interventions — tumor necrosis factor-alpha, CNGRC fusion protein, human; Doxorubicin

STUDY DESIGN:
Intervention Model Description: Dose-escalating study
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: NGR-hTNF; Drug: Doxorubicin

INTERVENTIONS:
Drug: NGR-hTNF — 0.2, 0.4, 0.8 and 1.6 μg/m²as 60-minute intravenous infusion every 3 weeks
Drug: Doxorubicin — 75 mg/m² intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)

SUMMARY:
The main objective of the trial is to document the safety of the combination (escalation doses of NGR-hTNF, from 0.2 mcg/sqm to 1.6 mcg/sqm , with a fixed dose of doxorubicin, 75 mg/sqm). Safety will be established by clinical and laboratory assessment according to National Cancer Institute Common Toxicity Criteria (NCI-CTC ).

DETAILED DESCRIPTION:
This is a phase IB, open-label, non-randomized, dose-escalation study that will be conducted in sequential cohorts of patients. Three patients per each cohort are planned.

Patients, with advanced or metastatic solid tumor previously treated with a non cumulative dose of doxorubicin (<300 mg/sqm in order to allow an adequate number of cycles) or chemotherapy naïve will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old with proven advanced or metastatic solid tumor not amenable to any clinical improvement by current standard treatments and previously treated with a non cumulative dose of anthracyclines (<300 mg/sqm) or chemotherapy naïve.
* Life expectancy more than 3 months.
* ECOG performance status 0 - 2.
* Normal cardiac function (left ventricular ejection fraction [LVEF] ≥55%) and absence of uncontrolled hypertension.
* Absence of any conditions involving hypervolemia and its consequences.
* Adequate baseline bone marrow, hepatic and renal function, defined as follows:

Neutrophils > 1.5 x 10^9/L and platelets >100 x 10^9/L Bilirubin < 1.5 x ULN AST and/or ALT < 2 x ULN Serum creatinine < 1.5 x ULN

* Patients may have had prior therapy providing the following conditions are met:

  * Chemo, radio, hormonal, immuno or anti-vascular therapy: wash-out period of 28 days.
  * Surgery: wash-out period of 14 days.
* Patients must give written informed consent to participate in the study.

Exclusion Criteria:

* Concurrent anticancer therapy
* Patients must not receive any other investigational agents while on study
* Patients with a LVEF <55%
* New York Heart Association class III or IV cardiac disease
* Acute angina
* Patients with myocardial infarction within the last six (6) months
* Patient with significant peripheral vascular disease
* Thrombosis of main portal vein
* Previous signs of severe toxicity doxorubicin related
* Previous signs of cardiotoxicity doxorubicin related
* Patients previously treated with a cumulative dosage of anthracyclines ≥300 mg/m^2
* Clinical signs of CNS involvement
* Patients with active or uncontrolled systemic disease/infections or with serious illness or medical conditions, which is incompatible with the protocol
* Known hypersensitivity/allergic reaction to human albumin preparations or to any of the excipients
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol
* Pregnancy or lactation. Patients - both males and females - with reproductive potential (i.e. menopausal for less than 1-year and not surgically sterilized) must practice effective contraceptive measures throughout the study. Women of child-bearing potential must provide a negative pregnancy test (serum or urine) within 14 days prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-02-28; Primary Completion 2007-05-08 (Actual); Study Completion 2007-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Federico Caligaris Cappio, MD, Principal Investigator — Fondazione San Raffaele del Monte Tabor
Locations (4):
- Italy (3):
  - Istituto Clinico Humanitas, Rozzano, Milan
  - Azienda Ospedaliera Universitaria "San Martino", Genova
  - Fondazione San Raffaele del Monte Tabor, Milan
- University Medical Centre, Nijmegen, Nijmegen, Netherlands

REFERENCES:
- [Background] Sacchi A, Gasparri A, Gallo-Stampino C, Toma S, Curnis F, Corti A. Synergistic antitumor activity of cisplatin, paclitaxel, and gemcitabine with tumor vasculature-targeted tumor necrosis factor-alpha. Clin Cancer Res. 2006 Jan 1;12(1):175-82. doi: 10.1158/1078-0432.CCR-05-1147. PMID 16397040

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Period: 28 February 2006 (first enrollment); 8 May 2007 (last completed). 3 investigational centres in Italy and 1 in Netherlands.
Pre-assignment Details: Screening details:
  Planned sample size: 20-25 patients; Patients screened n.: 15; Patients screening failure n.: 0.
Groups:
- Cohort 1: NGR-hTNF 0.2 μg/m^2+ Doxorubicin 60 mg/m^2: NGR-hTNF: 0.2 μg/m^2 as 60-minute intravenous infusion every 3 weeks
  Doxorubicin: 60 mg/m^2 intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
- Cohort 2: NGR-hTNF 0.2 μg/m^2+ Doxorubicin 75 mg/m^2: NGR-hTNF: 0.2 μg/m^2 as 60-minute intravenous infusion every 3 weeks
  Doxorubicin: 75 mg/m^2 intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
- Cohort 3: NGR-hTNF 0.4 μg/m^2+ Doxorubicin 75 mg/m^2: NGR-hTNF: 0.4 μg/m^2 as 60-minute intravenous infusion every 3 weeks
  Doxorubicin: 75 mg/m^2 intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
- Cohort 4: NGR-hTNF 0.8 μg/m^2+ Doxorubicin 75 mg/m^2: NGR-hTNF: 0.8 μg/m^2 as 60-minute intravenous infusion every 3 weeks
  Doxorubicin: 75 mg/m^2 intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
- Cohort 5: NGR-hTNF 1.6 μg/m^2+ Doxorubicin 75 mg/m^2: NGR-hTNF: 1.6 μg/m^2 as 60-minute intravenous infusion every 3 weeks
  Doxorubicin: 75 mg/m^2 intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
Period: Overall Study
Arm/Group | Cohort 1: NGR-hTNF 0.2 μg/m^2+ Doxorubicin 60 mg/m^2 | Cohort 2: NGR-hTNF 0.2 μg/m^2+ Doxorubicin 75 mg/m^2 | Cohort 3: NGR-hTNF 0.4 μg/m^2+ Doxorubicin 75 mg/m^2 | Cohort 4: NGR-hTNF 0.8 μg/m^2+ Doxorubicin 75 mg/m^2 | Cohort 5: NGR-hTNF 1.6 μg/m^2+ Doxorubicin 75 mg/m^2
Started | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: NGRhTNF 0.2 μg/m^2+ Doxorubicin 60 mg/m^2: NGR-hTNF: 0.2 μg/m^2as 60-minute intravenous infusion every 3 weeks
  Doxorubicin: 60 mg/m^2 intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
- Cohort 2: NGRhTNF 0.2 μg/m^2+ Doxorubicin 75 mg/m^2: NGR-hTNF: 0.2 μg/m^2as 60-minute intravenous infusion every 3 weeks
  Doxorubicin: 75 mg/m^2 intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
- Cohort 3: NGRhTNF 0.4 μg/m^2+ Doxorubicin 75 mg/m^2: NGR-hTNF: 0.4 μg/m^2as 60-minute intravenous infusion every 3 weeks
  Doxorubicin: 75 mg/m^2 intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
- Cohort 4: NGRhTNF 0.8 μg/m^2+ Doxorubicin 75 mg/m^2: NGR-hTNF: 0.8 μg/m^2as 60-minute intravenous infusion every 3 weeks
  Doxorubicin: 75 mg/m^2 intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
- Cohort 5: NGRhTNF 1.6 μg/m^2+ Doxorubicin 75 mg/m^2: NGR-hTNF: 1.6 μg/m^2as 60-minute intravenous infusion every 3 weeks
  Doxorubicin: 75 mg/m^2 intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
- Total: Total of all reporting groups
Arm/Group | Cohort 1: NGRhTNF 0.2 μg/m^2+ Doxorubicin 60 mg/m^2 | Cohort 2: NGRhTNF 0.2 μg/m^2+ Doxorubicin 75 mg/m^2 | Cohort 3: NGRhTNF 0.4 μg/m^2+ Doxorubicin 75 mg/m^2 | Cohort 4: NGRhTNF 0.8 μg/m^2+ Doxorubicin 75 mg/m^2 | Cohort 5: NGRhTNF 1.6 μg/m^2+ Doxorubicin 75 mg/m^2 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 2 | 3 | 2 | 13
  >=65 years | 0 | 0 | 1 | 0 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 0 | 1 | 0 | 5
  Male | 1 | 1 | 3 | 2 | 3 | 10
Region of Enrollment [Number; unit: participants]
  Netherlands | 1 | 2 | 0 | 1 | 1 | 5
  Italy | 2 | 1 | 3 | 2 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events From Escalating Doses of NGR-hTNF in Combination With a Fixed Dose of Doxorubicin
Description: An Adverse Event (AE) is any untoward medical occurrence or experience in a patient or clinical investigation subject treated administered a pharmaceutical product and which does not necessarily have to have a casual relationship with this treatment. An adverse event (AE) can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Through study completion, an average of 1 year
Measure: Number; unit: Adverse event
Groups:
- Cohort 1: NGRhTNF 0.2 μg/m^2+ Doxorubicin 60 mg/m^2: NGR-hTNF: 0.2 μg/m^2 as 60-minute intravenous infusion every 3 weeks Doxorubicin: 60 mg/m^2 intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
- Cohort 2: NGRhTNF 0.2 μg/m^2+ Doxorubicin 75 mg/m^2: NGR-hTNF: 0.2 μg/m^2 as 60-minute intravenous infusion every 3 weeks Doxorubicin: 75 mg/m^2 intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
- Cohort 3: NGR-hTNF 0.4 μg/m^2+ Doxorubicin 75 mg/m^2: NGR-hTNF: 0.4 μg/m^2 as 60-minute intravenous infusion every 3 weeks Doxorubicin:75 mg/m^2 intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
- Cohort 5:NGR-hTNF 1.6 μg/m^2+ Doxorubicin 75 mg/m^2: NGR-hTNF: 1.6 μg/m^2 as 60-minute intravenous infusion every 3 weeks Doxorubicin: 75 mg/m^2 intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
Arm/Group | Cohort 1: NGRhTNF 0.2 μg/m^2+ Doxorubicin 60 mg/m^2 | Cohort 2: NGRhTNF 0.2 μg/m^2+ Doxorubicin 75 mg/m^2 | Cohort 3: NGR-hTNF 0.4 μg/m^2+ Doxorubicin 75 mg/m^2 | Cohort 4: NGR-hTNF 0.8 μg/m^2+ Doxorubicin 75 mg/m^2 | Cohort 5:NGR-hTNF 1.6 μg/m^2+ Doxorubicin 75 mg/m^2
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3
Adverse event | 59 | 142 | 67 | 101 | 124
Statistical Analysis 1: Comparison: Cohort 1: NGRhTNF 0.2 μg/m^2+ Doxorubicin 60 mg/m^2 vs Cohort 2: NGRhTNF 0.2 μg/m^2+ Doxorubicin 75 mg/m^2 vs Cohort 3: NGR-hTNF 0.4 μg/m^2+ Doxorubicin 75 mg/m^2 vs Cohort 4: NGR-hTNF 0.8 μg/m^2+ Doxorubicin 75 mg/m^2 vs Cohort 5:NGR-hTNF 1.6 μg/m^2+ Doxorubicin 75 mg/m^2; All data regarding safety were registered and analyzed by descriptive analyses. Summary table were generated to document the safety; Test type: Other; MDT = 1.6; at least 3 patients per cohort had to be enrolled with expansion to 6 in presence of Dose Limiting Toxicity(DLT) (stop escalation if 2 or more DLTs at the same dose level). With a projection to achieve the highest level of NGR-hTNF, without significative toxicity (1.6 μg/m2) a planned sample of 20-25 patients was expected. DLTs were defined as: any severe toxicity clearly related to the administration of NGR-hTNF. The patient was defined assessable, according to the standard analysis, if he/she received at least one infusion of the investigational product. Maximal Tollerated Dose (MTD) was defined as the dose which produces DLTs in 2 or more patients out of 6 and will be recommended for phase II trials

2. Secondary Outcome: Pharmacokinetic Profiles of NGR-hTNF Administrated in Combination With Doxorubicin (Cmax)
Description: Pharmacokinetic profiles of NGR-hTNF and doxorubicin was conducted in 4 sequential cohorts of patients (Three patients per each cohort were planned). The first 3 patients of the first cohort were treated with 0.2 μg/m2 of NGR-hTNF in combination with a suboptimal dose (minus 20%) of doxorubicin (60 mg/m2).Following 4 cohorts were treated with escalating dose of NGR-hTNF (0.2, 0.4, 0.8 and 1.6 μg/m2) in combination with a standard dose of doxorubicin (75 mg/m2):
Time Frame: prior to infusion and 15', 30', 60', 90', 120', 134' [1 minute before the end of doxorubicin administration], 180', 240', 360' minutes
Population: Pharmacokinetic of NGR-hTNF was conducted in 5 sequential cohorts of patients, 3 patients per each cohort were planned). All the patients treated on Cycle 1 were still in the study on Cycle2. On Cycle3 twelve out of fifteen patients were still in the study. Subjects no more included in the study were 1 patient in cohort 1 and 2 patients in cohort 5
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Cohort 2: NGR-hTNF 0.2 μg/m^2 + Doxorubicin 75 mg/m^2: NGR-hTNF: 0.2 μg/m^2 as 60-minute intravenous infusion every 3 weeks
  Doxorubicin: 75 mg/m² intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
- Cohort 3: NGR-hTNF 0.4 μg/m^2 + Doxorubicin 75 mg/m^2: NGR-hTNF: 0.4 μg/m^2 as 60- minute intravenous infusion every 3 weeks
  Doxorubicin: 75 mg/m^2 intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
- Cohort 4: NGR-hTNF 0.8 μg/m^2 + Doxorubicin 75 mg/m^2: NGR-hTNF: 0.8 μg/m^2 as 60-minute intravenous infusion every 3 weeks
  Doxorubicin: 75 mg/m^2 intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
- Cohort 5: NGR-hTNF 1.6 μg/m^2 + Doxorubicin 75 mg/m^2: NGR-hTNF: 1.6 μg/m^2 as 60-minute intravenous infusion every 3 weeks
  Doxorubicin: 75 mg/m^2 intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
Arm/Group | Cohort 1: NGR-hTNF 0.2 μg/m^2+ Doxorubicin 60 mg/m^2 | Cohort 2: NGR-hTNF 0.2 μg/m^2 + Doxorubicin 75 mg/m^2 | Cohort 3: NGR-hTNF 0.4 μg/m^2 + Doxorubicin 75 mg/m^2 | Cohort 4: NGR-hTNF 0.8 μg/m^2 + Doxorubicin 75 mg/m^2 | Cohort 5: NGR-hTNF 1.6 μg/m^2 + Doxorubicin 75 mg/m^2
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3
pg/mL
  Cycle1_Cmax NGR-hTNF | 2.22 (0.58) | 1.82 (0.90) | 4.44 (1.70) | 8.10 (1.50) | 15.7 (8.34)
  Cycle2_Cmax NGR-hTNF | 3.10 (1.54) | 2.31 (1.69) | 2.74 (2.94) | 18.0 (15.6) | 34.4 (22.5)
  Cycle3_Cmax NGR-hTNF: number analyzed (Participants) | 2 | 3 | 3 | 3 | 1
  Cycle3_Cmax NGR-hTNF | 2.28 (0.21) | 3.04 (2.14) | 8.91 (8.70) | 11.2 (5.90) | 25.4

3. Secondary Outcome: Pharmacokinetic Profiles of NGR-hTNF Administrated in Combination With Doxorubicin (Tmax)
Description: as for outcome 2
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Groups:
- Cohort 2: NGR-hTNF 0.2 μg/m^2 + Doxorubicin 75 mg/m^2: NGR-hTNF: 0.2 μg/m^2 as 60-minute intravenous infusion every 3 weeks
  Doxorubicin: 75 mg/m^2 intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
Arm/Group | Cohort 1: NGR-hTNF 0.2 μg/m^2+ Doxorubicin 60 mg/m^2 | Cohort 2: NGR-hTNF 0.2 μg/m^2 + Doxorubicin 75 mg/m^2 | Cohort 3: NGR-hTNF 0.4 μg/m^2+ Doxorubicin 75 mg/m^2 | Cohort 4: NGR-hTNF 0.8 μg/m^2+ Doxorubicin 75 mg/m^2 | Cohort 5: NGR-hTNF 1.6 μg/m^2 + Doxorubicin 75 mg/m^2
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3
h
  Cycle1_tmax_NGR-hTNF | 0.25 (0.00) | 2.50 (3.04) | 2.50 (3.04) | 0.78 (0.39) | 2.83 (3.18)
  Cycle2_tmax NGR-hTNF | 0.87 (0.29) | 2.42 (3.13) | 1.03 (0.46) | 0.75 (0.35) | 0.83 (0.29)
  Cycle3_tmax NGR-hTNF: number analyzed (Participants) | 2 | 3 | 3 | 3 | 1
  Cycle3_tmax NGR-hTNF | 1.04 (0.057) | 4.08 (3.32) | 0.83 (0.29) | 0.67 (0.29) | 6.00

4. Secondary Outcome: Pharmacokinetic Profiles of NGR-hTNF Administrated in Combination With Doxorubicin (AUC0-t(Last))
Description: as for outcome 2
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg⋅h/mL
Groups:
- Cohort 1: NGR-hTNF 0.2 μg/m^2 + Doxorubicin 60 mg/m^2: NGR-hTNF: 0.2 μg/m^2 as 60-minute intravenous infusion every 3 weeks
  Doxorubicin: 60 mg/m^2 intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
- Cohort 3: NGR-hTNF 0.4 μg/m^2 + Doxorubicin 75 mg/m^2: NGR-hTNF: 0.4 μg/m^2 as 60-minute intravenous infusion every 3 weeks
  Doxorubicin: 75 mg/m^2 intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
Arm/Group | Cohort 1: NGR-hTNF 0.2 μg/m^2 + Doxorubicin 60 mg/m^2 | Cohort 2: NGR-hTNF 0.2 μg/m^2 + Doxorubicin 75 mg/m^2 | Cohort 3: NGR-hTNF 0.4 μg/m^2 + Doxorubicin 75 mg/m^2 | Cohort 4: NGR-hTNF 0.8 μg/m^2 + Doxorubicin 75 mg/m^2 | Cohort 5: NGR-hTNF 1.6 μg/m^2 + Doxorubicin 75 mg/m^2
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3
pg⋅h/mL
  Cycle1_AUC0-t(last)_NGR-hTNF | 1.94 (0.27) | 1.99 (1.42) | 11.8 (4.13) | 12.0 (0.70) | 25.7 (19.4)
  Cycle2_AUC0-t(last)_ NGR-hTNF | 7.84 (7.06) | 2.74 (1.63) | 4.53 (5.95) | 20.5 (13.0) | 46.4 (28.9)
  Cycle3_AUC0-t(last)_NGR-hTNF: number analyzed (Participants) | 2 | 3 | 3 | 3 | 1
  Cycle3_AUC0-t(last)_NGR-hTNF | 4.35 (0.40) | 2.71 (1.11) | 10.6 (7.13) | 18.2 (7.49) | 64.0

5. Secondary Outcome: sTNFRs and Anti-NGR-hTNF Antibody Plasma Levels (Emax)
Description: Pharmacodynamic calculations for sTNF-R1 and sTNF-R2 were performed on the plasma concentrations from which the baseline concentrations were subtracted (i.e. on positive and negative values). At all doses, Emax, i.e. the maximal stimulatory effect, and tmax were estimated as the coordinates of the highest point of the plasma profile (y, x axis, respectively)
Time Frame: as for outcome 2
Population: Pharmacodynamic of NGR-hTNF was conducted in 5 sequential cohorts of patients, 3 patients per each cohort were planned). All the patients treated on Cycle 1 were still in the study on Cycle2. On Cycle3 twelve out of fifteen patients were still in the study. Subjects no more included in the study were 1 patient in cohort 1 and 2 patients in cohort 5
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Cohort 2: NGR-hTNF 0.2 μg/m^2 + Doxorubicin 75mg/m^2: NGR-hTNF: 0.2 μg/m^2 as 60-minute intravenous infusion every 3 weeks
  Doxorubicin: 75 mg/m^2 intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
- Cohort 3: NGR-hTNF 0.4 μg/m^2 + Doxorubicin 75 mg/m^2: NGR-hTNF: 0.2, 0.4, 0.8 and 1.6 μg//m^2 as 60-minute intravenous infusion every 3 weeks
  Doxorubicin: 75 mg/m^2 intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
- Cohort 4: NGR-hTNF 0.8 μg/m^2+ Doxorubicin 75mg/m^2: NGR-hTNF: 0.8 μg/m^2 as 60-minute intravenous infusion every 3 weeks
  Doxorubicin: 75 mg/m^2 intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
- Cohort 5: NGR-hTNF 1.6 μg/m^2 + Doxorubicin 75mg/m^2: NGR-hTNF: 1.6 μg/m^2as 60-minute intravenous infusion every 3 weeks
  Doxorubicin: 75 mg/m^2 intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
Arm/Group | Cohort 1: NGR-hTNF 0.2 μg/m^2 + Doxorubicin 60 mg/m^2 | Cohort 2: NGR-hTNF 0.2 μg/m^2 + Doxorubicin 75mg/m^2 | Cohort 3: NGR-hTNF 0.4 μg/m^2 + Doxorubicin 75 mg/m^2 | Cohort 4: NGR-hTNF 0.8 μg/m^2+ Doxorubicin 75mg/m^2 | Cohort 5: NGR-hTNF 1.6 μg/m^2 + Doxorubicin 75mg/m^2
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3
ng/mL
  Cycle 1_Emax sTNF-R1 | 0.34 (0.08) | -0.19 (0.60) | 0.21 (0.26) | 0.59 (0.46) | 1.64 (0.69)
  Cycle 1_Emax sTNF-R2 | 0.01 (0.07) | 0.26 (0.10) | 0.13 (0.14) | 0.56 (0.40) | 2.23 (0.80)
  Cycle 2_Emax sTNF-R1 | 0.49 (0.11) | 0.21 (0.31) | 0.45 (0.33) | 0.69 (0.46) | 1.21 (0.80)
  Cycle 2_Emax sTNF-R2 | 0.31 (0.40) | -0.12 (0.25) | 0.33 (0.21) | 1.31 (0.79) | 2.62 (1.64)
  Cycle 3_Emax sTNF-R1: number analyzed (Participants) | 2 | 3 | 3 | 3 | 1
  Cycle 3_Emax sTNF-R1 | 0.44 (0.13) | 0.51 (0.48) | 0.38 (0.13) | 0.84 (0.11) | 0.88 (1)
  Cycle 3_Emax sTNF-R2: number analyzed (Participants) | 2 | 3 | 3 | 3 | 1
  Cycle 3_Emax sTNF-R2 | 0.11 (0.04) | -0.13 (0.12) | 0.37 (0.17) | 1.10 (0.24) | 1.44 (1)

6. Secondary Outcome: sTNFRs and Anti-NGR-hTNF Antibody Plasma Levels (Tmax)
Description: as for outcome 5
Time Frame: as for outcome 2
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: h
Groups:
- Cohort 3: NGR-hTNF 0.4 μg/m^2 + Doxorubicin 75mg/m^2: NGR-hTNF: 0.4 μg/m^2 as 60-minute intravenous infusion every 3 weeks
  Doxorubicin: 75 mg/m^2 intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
- Cohort 4: NGR-hTNF 0.8 μg/m^2 + Doxorubicin 75mg/m^2: NGR-hTNF: 0.8 μg/m^2 as 60-minute intravenous infusion every 3 weeks
  Doxorubicin: 75 mg//m^2 intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
- Cohort 5: NGR-hTNF 1.6 μg/m^2+ Doxorubicin 75mg/m^2: NGR-hTNF: 1.6 μg/m^2 as 60-minute intravenous infusion every 3 weeks
  Doxorubicin: 75 mg/m^2 intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
Arm/Group | Cohort 1: NGR-hTNF 0.2 μg/m^2 + Doxorubicin 60 mg/m^2 | Cohort 2: NGR-hTNF 0.2 μg/m^2 + Doxorubicin 75 mg/m^2 | Cohort 3: NGR-hTNF 0.4 μg/m^2 + Doxorubicin 75mg/m^2 | Cohort 4: NGR-hTNF 0.8 μg/m^2 + Doxorubicin 75mg/m^2 | Cohort 5: NGR-hTNF 1.6 μg/m^2+ Doxorubicin 75mg/m^2
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3
h
  Cycle 1_Tmax sTNF-R1 | 5.47 (1.17) | 2.17 (3.32) | 4.33 (2.89) | 3.78 (3.15) | 2.83 (3.18)
  Cycle 1_Tmax sTNF-R2 | 3.19 (3.00) | 0.25 (0.00) | 3.67 (2.52) | 1.78 (0.32) | 2.83 (3.18)
  Cycle 2_Tmax sTNF-R1 | 4.71 (1.25) | 6.00 (0.00) | 4.33 (2.89) | 4.12 (2.67) | 1.17 (0.29)
  Cycle 2_Tmax sTNF-R2 | 4.71 (1.25) | 1.42 (1.42) | 3.67 (2.52) | 1.50 (0.71) | 1.17 (0.29)
  Cycle 3_Tmax sTNF-R1: number analyzed (Participants) | 3 | 3 | 3 | 3 | 1
  Cycle 3_Tmax sTNF-R1 | 6.09 (0.12) | 2.33 (3.18) | 5.33 (1.16) | 1.84 (1.04) | 6.00
  Cycle 3_Tmax sTNF-R2: number analyzed (Participants) | 2 | 3 | 3 | 3 | 1
  Cycle 3_Tmax sTNF-R2 | 6.09 (0.12) | 2.33 (3.18) | 3.50 (2.78) | 1.18 (0.31) | 1.00

7. Secondary Outcome: sTNFRs and Anti-NGR-hTNF Antibody Plasma Levels (ARC)
Description: as for outcome 5
Time Frame: as for outcome 2
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng⋅h/mL
Groups:
- Cohort 2: NGR-hTNF 0.2μg/m^2 + Doxorubicin 75mg/m^2: NGR-hTNF: 0.2 μg/m^2 as 60-minute intravenous infusion every 3 weeks
  Doxorubicin: 75 mg/m^2 intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
- Cohort 4: NGR-hTNF 0.8 μg/m^2 + Doxorubicin 75mg/m^2: NGR-hTNF: 0.8 μg/m^2 as 60-minute intravenous infusion every 3 weeks
  Doxorubicin: 75 mg/m^2 intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
- Cohort 5: NGR-hTNF 1.6 μg/m^2+ Doxorubicin 75mg/m^2: NGR-hTNF: 1.6 μg//m^2 as 60-minute intravenous infusion every 3 weeks
  Doxorubicin: 75 mg/m^2intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
Arm/Group | Cohort 1: NGR-hTNF 0.2 μg/m^2 + Doxorubicin 60 mg/m^2 | Cohort 2: NGR-hTNF 0.2μg/m^2 + Doxorubicin 75mg/m^2 | Cohort 3: NGR-hTNF 0.4 μg/m^2 + Doxorubicin 75mg/m^2 | Cohort 4: NGR-hTNF 0.8 μg/m^2 + Doxorubicin 75mg/m^2 | Cohort 5: NGR-hTNF 1.6 μg/m^2+ Doxorubicin 75mg/m^2
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3
ng⋅h/mL
  Cycle 1_ARC sTNF-R1 | 0.1 (0.24) | -3.52 (3.71) | -0.64 (0.86) | 2.11 (1.72) | 3.38 (0.81)
  Cycle 1_ARC sTNF-R2 | -1.04 (1.12) | -1.58 (1.17) | -1.36 (2.22) | 2.10 (1.41) | 6.08 (3.40)
  Cycle 2_ARC sTNF-R1 | 0.75 (0.27) | -0.57 (0.58) | 0.74 (1.38) | 1.76 (1.01) | 3.38 (2.85)
  Cycle 2_ARC sTNF-R2 | 0.35 (1.16) | -2.89 (0.28) | 0.28 (1.03) | 2.95 (0.04) | 9.08 (7.17)
  Cycle 3_ARC sTNF-R1: number analyzed (Participants) | 2 | 3 | 3 | 3 | 1
  Cycle 3_ARC sTNF-R1 | 0.32 (0.29) | 0.11 (1.56) | 0.85 (0.37) | 2.49 (0.66) | 2.55
  Cycle 3_ARC sTNF-R2: number analyzed (Participants) | 2 | 3 | 3 | 3 | 1
  Cycle 3_ARC sTNF-R2 | -1.08 (0.09) | -3.30 (2.06) | 0.61 (0.34) | 3.25 (1.00) | 5.58

8. Secondary Outcome: sTNFRs and Anti-NGR-hTNF Antibody Plasma Levels (Eav)
Description: as for outcome 5
Time Frame: as for outcome 2
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Cohort 3: NGR-hTNF 0.4 μg/m^2 + Doxorubicin 75mg/m^2: NGR-hTNF: 0.4 μg/m^2as 60-minute intravenous infusion every 3 weeks
  Doxorubicin: 75 mg/m^2 intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
- Cohort 5: NGR-hTNF 1.6 μg/m^2 + Doxorubicin 75mg/m^2: NGR-hTNF: 1.6 μg/m^2 as 60-minute intravenous infusion every 3 weeks
  Doxorubicin: 75 mg/m^2 intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
Arm/Group | Cohort 1: NGR-hTNF 0.2 μg/m^2 + Doxorubicin 60 mg/m^2 | Cohort 2: NGR-hTNF 0.2 μg/m^2 + Doxorubicin 75mg/m^2 | Cohort 3: NGR-hTNF 0.4 μg/m^2 + Doxorubicin 75mg/m^2 | Cohort 4: NGR-hTNF 0.8 μg/m^2 + Doxorubicin 75mg/m^2 | Cohort 5: NGR-hTNF 1.6 μg/m^2 + Doxorubicin 75mg/m^2
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3
ng/mL
  Cycle 1_Eav sTNF-R1 | 0.02 (0.04) | -0.59 (0.62) | -0.11 (0.14) | 0.35 (0.29) | 0.56 (0.14)
  Cycle 1_Eav sTNF-R2 | -0.17 (0.19) | -0.26 (0.20) | -0.23 (0.37) | 0.35 (0.24) | 1.01 (0.57)
  Cycle 2_Eav sTNF-R1 | 0.13 (0.05) | -0.10 (0.10) | 0.12 (0.23) | 0.29 (0.17) | 0.56 (0.48)
  Cycle 2_Eav sTNF-R2 | 0.06 (0.19) | -0.48 (0.05) | 0.003 (0.17) | 0.49 (0.01) | 1.51 (1.20)
  Cycle 3_Eav sTNF-R1: number analyzed (Participants) | 2 | 3 | 3 | 3 | 1
  Cycle 3_Eav sTNF-R1 | 0.05 (0.05) | 0.02 (0.26) | 0.14 (0.06) | 0.42 (0.11) | 0.43
  Cycle 3_Eav sTNF-R2: number analyzed (Participants) | 2 | 3 | 3 | 3 | 1
  Cycle 3_Eav sTNF-R2 | -0.18 (0.02) | -0.55 (0.34) | 0.10 (0.06) | 0.54 (0.17) | 0.93

9. Secondary Outcome: To Evaluate Phenotype Analysis and Adaptative Immune Response
Time Frame: during the study
Population: No analysis was performed. No biopsy was preformed.
Groups:
- NGR-hTNF: 0.2, 0.4, 0.8 and 1.6 μg/m²as 60-minute Intravenous: NGR-hTNF: 0.2, 0.4, 0.8 and 1.6 μg/m²as 60-minute intravenous infusion every 3 weeks
  Doxorubicin: 75 mg/m² intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
Arm/Group | NGR-hTNF: 0.2, 0.4, 0.8 and 1.6 μg/m²as 60-minute Intravenous
Number analyzed (Participants) | 0

10. Secondary Outcome: Signs of Anticancer Activity by Standard Imaging or Clinically; When Possible Tumor Response Will be Documented According to RECIST Criteria
Description: Response to treatment was assessed on a set of target lesions(TL) chosen before the 1st treatment administration, the list of TL must be reported on the initial measurement form before the start of treatment. Lesions had to have clearly defined borders and initially were measured in at least one dimension, and had to be repeated at each evaluation of the disease by the same method. Sum of the longest diameter (LD) was calculated as the baseline sum LD Complete Response(CR): Disappearance of all TL Partial Response(PR): At least a 30% decrease in the sum of the LD of TL, taking as reference the base line sum LD Progressive Disease(PD): At least a 20% increase in the sum of LD of TL, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions Stable Disease (SD):Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started
Time Frame: after the first 2 cycles(Follow-up 2) of treatment and then every 2 cycles (Follow-up 4,6..). In case of detection of a complete or partial response, a confirmation assessment must be performed ≥ 4 weeks after the first documentation of the response.
Population: disease progression or until the start of another treatment
Measure: Number; unit: participants
Groups:
- Cohort 1: NGRhTNF 0.2 μg/m^2+ Doxorubicin 60 mg/m^2: NGR-hTNF: 0.2 μg/m^2 as 60-minute intravenous infusion every 3 weeks
  Doxorubicin: 60 mg/m² intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
- Cohort 2: NGRhTNF 0.2 μg/m^2+ Doxorubicin 75 mg/m^2: NGR-hTNF: 0.2 μg/m^2 as 60-minute intravenous infusion every 3 weeks
  Doxorubicin: 75 mg/m² intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
- Cohort 3: NGR-hTNF 0.4 μg/m^2+ Doxorubicin 75 mg/m^2: NGR-hTNF: 0.4 μg/m^2 as 60-minute intravenous infusion every 3 weeks
  Doxorubicin: 75 mg/m² intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
- Cohort 4: NGR-hTNF 0.8 μg/m^2+ Doxorubicin 75 mg/m^2: NGR-hTNF: 0.8 μg/m^2 as 60-minute intravenous infusion every 3 weeks
  Doxorubicin: 75 mg/m² intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
- Cohort 5: NGR-hTNF 1.6 μg/m^2+ Doxorubicin 75 mg/m^2: NGR-hTNF: 1.6 μg/m^2 as 60-minute intravenous infusion every 3 weeks
  Doxorubicin: 75 mg/m² intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
Arm/Group | Cohort 1: NGRhTNF 0.2 μg/m^2+ Doxorubicin 60 mg/m^2 | Cohort 2: NGRhTNF 0.2 μg/m^2+ Doxorubicin 75 mg/m^2 | Cohort 3: NGR-hTNF 0.4 μg/m^2+ Doxorubicin 75 mg/m^2 | Cohort 4: NGR-hTNF 0.8 μg/m^2+ Doxorubicin 75 mg/m^2 | Cohort 5: NGR-hTNF 1.6 μg/m^2+ Doxorubicin 75 mg/m^2
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3
participants
  N. of Stable Disease_follow-up 2 | 2 | 3 | 3 | 2 | 3
  N. of Progression Disease_follow-up 2 | 1 | 0 | 0 | 0 | 0
  N. of Partial Response follow-up 2 | 0 | 0 | 0 | 1 | 0
  N. of Stable Disease_follow-up 4: number analyzed (Participants) | 2 | 3 | 2 | 3 | 1
  N. of Stable Disease_follow-up 4 | 1 | 2 | 1 | 2 | 1
  N. of Progression Disease_follow-up 4: number analyzed (Participants) | 2 | 3 | 2 | 3 | 1
  N. of Progression Disease_follow-up 4 | 1 | 1 | 1 | 0 | 0
  N. of Partial Response follow-up 4: number analyzed (Participants) | 2 | 3 | 2 | 3 | 1
  N. of Partial Response follow-up 4 | 0 | 0 | 0 | 1 | 0
  N. of Stable Disease_follow-up 6: number analyzed (Participants) | 1 | 2 | 1 | 3 | 1
  N. of Stable Disease_follow-up 6 | 1 | 1 | 0 | 2 | 1
  N. of Progression Disease_follow-up 6: number analyzed (Participants) | 1 | 2 | 1 | 3 | 1
  N. of Progression Disease_follow-up 6 | 0 | 0 | 1 | 0 | 0
  N. of Partial Response follow-up 6: number analyzed (Participants) | 1 | 2 | 1 | 3 | 1
  N. of Partial Response follow-up 6 | 0 | 1 | 0 | 1 | 0
  N. of Stable Disease_follow-up 8: number analyzed (Participants) | 0 | 2 | 0 | 3 | 0
  N. of Stable Disease_follow-up 8 |  | 1 |  | 1 |
  N. of Progression Disease_follow-up 8: number analyzed (Participants) | 0 | 2 | 0 | 3 | 0
  N. of Progression Disease_follow-up 8 |  | 1 |  | 2 |
  N. of Partial Response follow-up 8: number analyzed (Participants) | 0 | 2 | 0 | 3 | 0
  N. of Partial Response follow-up 8 |  | 0 |  | 0 |

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 1 year
Groups:
- Cohort 5: NGR-hTNF: 1.6 μg/m^2 + Doxorubicin 75 mg/m^2: NGR-hTNF: 1.6 μg/m^2 as 60-minute intravenous infusion every 3 weeks
  Doxorubicin: 75 mg/m² intravenous infusion over 15 minutes (starting 1 hour after the end of NGR-hTNF infusion)
Arm/Group | Cohort 1: NGRhTNF 0.2 μg/m^2+ Doxorubicin 60 mg/m^2 | Cohort 2: NGRhTNF 0.2 μg/m^2+ Doxorubicin 75 mg/m^2 | Cohort 3: NGR-hTNF 0.4 μg/m^2+ Doxorubicin 75 mg/m^2 | Cohort 4: NGR-hTNF 0.8 μg/m^2+ Doxorubicin 75 mg/m^2 | Cohort 5: NGR-hTNF: 1.6 μg/m^2 + Doxorubicin 75 mg/m^2
All-Cause Mortality (participants affected / at risk) | 2/3 | 1/3 | 2/3 | 0/3 | 2/3
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 2/3 | 3/3 | 1/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: NGRhTNF 0.2 μg/m^2+ Doxorubicin 60 mg/m^2 (N=3) | Cohort 2: NGRhTNF 0.2 μg/m^2+ Doxorubicin 75 mg/m^2 (N=3) | Cohort 3: NGR-hTNF 0.4 μg/m^2+ Doxorubicin 75 mg/m^2 (N=3) | Cohort 4: NGR-hTNF 0.8 μg/m^2+ Doxorubicin 75 mg/m^2 (N=3) | Cohort 5: NGR-hTNF: 1.6 μg/m^2 + Doxorubicin 75 mg/m^2 (N=3)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: NGRhTNF 0.2 μg/m^2+ Doxorubicin 60 mg/m^2 (N=3) | Cohort 2: NGRhTNF 0.2 μg/m^2+ Doxorubicin 75 mg/m^2 (N=3) | Cohort 3: NGR-hTNF 0.4 μg/m^2+ Doxorubicin 75 mg/m^2 (N=3) | Cohort 4: NGR-hTNF 0.8 μg/m^2+ Doxorubicin 75 mg/m^2 (N=3) | Cohort 5: NGR-hTNF: 1.6 μg/m^2 + Doxorubicin 75 mg/m^2 (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (5) | 2 (4) | 3 (10) | 2 (10)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (9) | 3 (12) | 3 (14) | 3 (10)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 1 (1) | 2 (16) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 2 (5) | 2 (8) | 3 (12) | 3 (18) | 3 (10)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 0 (0)
Asystole (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Mitral valve sclerosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abnormal sensation in eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dry eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 1 (8) | 0 (0) | 0 (0) | 2 (4)
Aptyalism (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (2) | 2 (7)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 1 (2)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (12) | 3 (9) | 1 (1) | 2 (5) | 2 (4)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus ani (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Teething (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (3) | 1 (3) | 0 (0) | 2 (2) | 3 (7)
Asthenia (General disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 1 (1) | 2 (4) | 2 (6) | 3 (5)
Fatigue (General disorders) | 2 (3) | 1 (5) | 0 (0) | 1 (2) | 2 (4)
Mucosal inflammation (General disorders) | 0 (0) | 1 (4) | 0 (0) | 1 (7) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (2) | 2 (6) | 0 (0) | 0 (0) | 2 (5)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mycosis fungoides (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Graft complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 1 (7) | 0 (0) | 0 (0) | 1 (2)
Troponin I (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (2) | 1 (3) | 0 (0) | 1 (1) | 2 (6)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pain in limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sacral pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Shoulder blade pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle tone abnormal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Neuropathic pain (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 2 (2) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mediastinal disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (5) | 0 (0) | 1 (2) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peely skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Red face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (14) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head cold (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Restless legs syndrome (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes